CLINICAL TRIAL: NCT01526538
Title: Improving Learning-based Treatment of Cocaine Dependence With Medication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Matthew Johnson, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21DA029823 (NIH)
Record Dates: First submitted 2012-01-30; First posted 2012-02-06 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: COCAINE-RELATED DISORDERS
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50 mg d-cycloserine (Experimental): active drug condition
  Interventions: Drug: d-cycloserine
- Sugar pill (Placebo Comparator): Inactive placebo
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: d-cycloserine — 50 mg d-cycloserine
  Arms: 50 mg d-cycloserine
Drug: sugar pill — placebo
  Arms: Sugar pill

SUMMARY:
This study will test the efficacy of d-cycloserine in enhancing response to learning-based treatment for cocaine dependence, specifically contingency management.

DETAILED DESCRIPTION:
Cocaine dependence is a public health problem with substantial morbidity, however no effective pharmacotherapy for cocaine dependence has been approved by the FDA. Unlike previous medication studies that have sought to pharmacologically reduce cocaine reinforcement, seeking or craving, this exploratory clinical trial will test d-cycloserine (DCS) for its ability to improve learning-based behavioral treatment of cocaine dependence. DCS is an NMDA partial agonist that has been shown to robustly improve learning in preclinical models, including extinction of cocaine conditioned place preference and blockade of cocaine reacquisition, and to improve extinction-learning based exposure therapy for multiple anxiety disorders. This Phase II clinical trial will investigate the pharmacological (DCS) enhancement of a behavioral treatment combining contingency management (CM) and novel home-environment exposure therapy sessions for cocaine dependence. High magnitude CM incentives will be used to promote the cocaine abstinence necessary for extinction in home-based exposure sessions. Participants will be randomized into 2 groups: 1. CM with placebo (CM+PL), and 2. CM with DCS (CM+DCS). For 19 days after group assignment, participants will report to the laboratory 3 times per week (Mon, Wed, Fri) to provide urine samples, receive contingent vouchers, and complete assessments of drug use, craving, mood, withdrawal, and quit self-efficacy. DCS (50 mg) or placebo will be administered on Mon, Wed and Fri study visits (at the end of the lab visit before returning to the home environment for exposure sessions during the time of DCS action). Follow-up visits will be conducted at 1 week, 1 month, and 3 months post-CM completion, during which time measures of drug use (self-reported and urinalysis), craving, mood, and withdrawal will be obtained. Comparison of continuous abstinence post-CM between the groups will be the primary outcome measure. During an initial laboratory session, a battery of learning/cognitive tasks will test for forms of learning/cognition enhanced by DCS that might contribute to the treatment effect. This project will test the efficacy of a novel intervention for cocaine dependence that was developed based on a known efficacious cocaine dependence treatment (CM), principles of extinction learning theory, and a medication shown to improve preclinical learning in general, including extinction of cocaine conditioning, and clinical learning-based exposure treatment of anxiety disorders. The study may indicate cost effective additions (home exposure sessions and DCS) to extend CM benefit after the removal of contingencies, and therefore may increase the dissemination of CM in community settings.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age (> 60 due to age-related effects on cognitive functioning)
* Satisfy DSM-IV criteria for cocaine dependence (primarily crack)
* Able to complete all study measures
* Currently seeking treatment for cocaine dependence

Exclusion Criteria:

* Meets DSM-IV criteria for dependence on a drug other than cocaine or nicotine (may meet abuse criteria for other drugs)
* Pregnant, breast feeding, or planning to become pregnant within 3 months
* If female, do not agree to use an effective means of birth control during the course of treatment (via phone screen)
* History of seizure disorder, severe hepatic impairment, porphyria, serious head trauma, dementia, or significant cognitive impairment
* Diagnosis of current major psychiatric disorder besides substance dependence or abuse
* Reported use of DCS in the past year
* Illiteracy, as will be determined during in-person screening
* Concurrently prescribed or using ethionamide or isoniazid (both used to treat tuberculosis)
* Positive urine result for opioids at screening interview

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Johnson MW, Bruner NR, Johnson PS, Silverman K, Berry MS. Randomized controlled trial of d-cycloserine in cocaine dependence: Effects on contingency management and cue-induced cocaine craving in a naturalistic setting. Exp Clin Psychopharmacol. 2020 Apr;28(2):157-168. doi: 10.1037/pha0000306. Epub 2019 Aug 1. PMID 31368770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 50 mg D-cycloserine | Sugar Pill
Started | 30 | 22
Completed | 21 | 18
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg D-cycloserine | Sugar Pill | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (5.3) | 52.1 (4.9) | 51.7 (5.1)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Urinalysis Benzoylecgonine (Cocaine Metabolite)(ng/ml)
Description: The primary outcome for this study will be post-treatment continuous abstinence, as assessed by urinalysis results
Time Frame: 1 month post-treatment
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 50 mg D-cycloserine | Sugar Pill
Number analyzed (Participants) | 22 | 18
ng/ml | 36.7 (7.7) | 32.4 (6.6)

2. Primary Outcome: Medication Side-effects
Description: self-report of medication side effects (Units of Measure is the count of specific reported effects)
Time Frame: 1 month post-treatment.
Measure: Number; unit: Adverse event reports
Groups:
- D-cycloserine: Study medication under investigation
- Control: Placebo (sugar pill)
Arm/Group | D-cycloserine | Control
Number analyzed (Participants) | 21 | 18
Adverse event reports | 0 | 0

3. Secondary Outcome: Learning Task by Itami and Uno
Time Frame: At the baseline laboratory visit
Measure: Mean (Standard Error); unit: % correct
Arm/Group | 50 mg D-cycloserine | Sugar Pill
Number analyzed (Participants) | 21 | 18
% correct | 81.5 (3.5) | 72.9 (4.4)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 50 mg D-cycloserine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No